CLINICAL TRIAL: NCT01078454
Title: A Randomized Phase III Trial of Melphalan and Dexamethasone (MDex) Versus Bortezomib, Melphalan and Dexamethasone (BMDex) for Untreated Patients With Systemic Light-Chain (AL) Amyloidosis Ineligible for Autologous Stem-Cell Transplantation
Brief Title: Melphalan and Dexamethasone With or Without Bortezomib in Treating Patients With Previously Untreated Systemic Light-Chain Amyloidosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02010; NCI-2011-02010 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E4A08 (Other: Eastern Cooperative Oncology Group (ECOG)); U10CA021115 (NIH)
Record Dates: First submitted 2010-02-27; First posted 2010-03-02 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Light Chain Deposition Disease; Primary Systemic Amyloidosis
Keywords: Melphalan; Dexamethasone; Bortezomib; Systemic Light-chain (AL) Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis | interventions — Melphalan; Dexamethasone; Calcium Dobesilate; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A (Mel-Dex) (Experimental): Patients receive melphalan 0.22 mg/kg orally (PO) and dexamethasone 40 mg PO on days 1-4 every 4 weeks. Treatment repeats every 4 weeks for up to 9 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: melphalan; Drug: dexamethasone
- ARM B (B-Mel-Dex) (Experimental): Patients receive melphalan 0.22 mg/kg PO and dexamethasone 40 mg PO on days 1-4 and bortezomib 1.3 mg/m^2 intravenously (IV) on days 1, 4, 8, and 11 every 4 weeks. Treatment repeats every 4 weeks for 2 cycles. Patients then receive melphalan PO and dexamethasone PO on days 1-4 and bortezomib IV on days 1, 8, 15, and 22 every 5 weeks. Treatment repeats every 5 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: melphalan; Drug: dexamethasone; Drug: bortezomib

INTERVENTIONS:
Drug: melphalan — Given PO
  Other Names: L-PAM; L-phenylalanine mustard; L-sarcolysin; Alkeran; NSC #8806
Drug: dexamethasone — Given PO
  Other Names: Decadron; Hexadrol; Dexameth; Dexone; DXM
Drug: bortezomib — Given IV
  Other Names: Velcade®; PS-341; MLN-341; LDP-341
  Arms: ARM B (B-Mel-Dex)

SUMMARY:
This randomized phase III trial is studying melphalan and dexamethasone to see how well they work with or without bortezomib in treating patients with previously untreated systemic amyloidosis. Drugs used in chemotherapy, such as melphalan and dexamethasone, work in different ways to stop the growth of plasma cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of plasma cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving melphalan together with dexamethasone is more effective with or without bortezomib in treating systemic amyloidosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare hematologic overall response (partial response [PR], very good PR, amyloid complete hematologic response [ACR], and stringent complete response [sCR]) after 3 courses of therapy in patients with previously untreated systemic light-chain amyloidosis treated with melphalan and dexamethasone with vs without bortezomib.

SECONDARY OBJECTIVES:

I. To evaluate the ACR rate after 3 courses of therapy and at completion of therapy.

II. To evaluate organ response rates after 3 courses of therapy and at 6, 9, and 12 months.

III. To evaluate treatment-related mortality.

IV. To evaluate toxicity.

V. To evaluate progression-free and overall survival.

VI. To evaluate PR or better at completion of therapy.

VII. To evaluate time to hematologic and organ response.

VIII. To evaluate the duration of hematologic and organ response.

IX. To assess quality of life (QOL) at baseline, at 3, 6, and 9 months during the therapy, at completion of therapy, and 3 and 6 months after therapy.

TERTIARY OBJECTIVES:

I. To determine the prognostic impact of t(11;14) translocation and cyclin D1 overexpression on response and overall survival.

II. (Correlative) To compare sCR rates and to determine the impact of sCR on the outcomes.

III. (Correlative) To perform a descriptive analysis of amyloid typing and proteomic composition of amyloid tissues.

OUTLINE: This is a multicenter study. Patients are stratified according to amyloid cardiac stage (stage I/II vs. better risk stage III) and are randomized to 1 of 2 treatment arms.

ARM A (Mel-Dex): Patients receive melphalan 0.22 mg/kg orally (PO) and dexamethasone 40 mg PO on days 1-4 every 4 weeks. Treatment repeats every 4 weeks for up to 9 courses in the absence of disease progression or unacceptable toxicity.

ARM B (B-Mel-Dex): Patients receive melphalan 0.22 mg/kg PO and dexamethasone 40 mg PO on days 1-4 and bortezomib 1.3 mg/m2 intravenously (IV) on days 1, 4, 8, and 11 every 4 weeks. Treatment repeats every 4 weeks for 2 cycles. Patients then receive melphalan PO and dexamethasone PO on days 1-4 and bortezomib IV on days 1, 8, 15, and 22 every 5 weeks. Treatment repeats every 5 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

Blood, urine, bone marrow, and fat samples may be collected periodically for laboratory analysis. Health-related quality of life is assessed periodically before, during, and after therapy. After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of systemic light-chain amyloidosis

  * Histologic diagnosis of disease must be confirmed by pathology (positive Congo red stain with green birefringence on polarized light microscopy)
  * Genetic testing must be negative for transthyretin mutations associated with hereditary amyloidosis (required in patients who are African-American or who present with peripheral neuropathy as the dominant organ involvement)
* Measurable disease, defined by >= 1 of the following:

  * Serum M-protein >= 1 g/dL by serum protein electrophoresis (SPEP)
  * Difference between involved and uninvolved free light chain be >4.0mg/dL provided the kappa to lambda free light chain (FLC) ratio is abnormal
* Symptomatic organ involvement* (heart, kidney, liver/gastrointestinal tract, peripheral nervous system, or soft tissue), defined as any of the following:

  * NOTE: *Carpal tunnel syndrome skin purpura or the presence of vascular amyloid on a bone marrow biopsy alone are not sufficient to meet criteria for "symptomatic organ involvement"
  * Renal involvement is defined as proteinuria (predominantly albumin) > 0.5 g/day by 24-hour urine collection
  * Cardiac involvement is defined as the presence of a mean left ventricular wall thickness of > 12 mm by echocardiogram in the absence of a history of hypertension or valvular heart disease or in the presence of unexplained low voltage (< 0.5 mV) by electrocardiogram
  * Hepatic involvement is defined as hepatomegaly or an alkaline phosphatase > 1.5 times upper limit of normal (ULN)
  * Peripheral nerve involvement is defined by clinical history or abnormal sensory and/or motor findings on neurologic exam
  * Gastrointestinal (GI) involvement is defined as gross GI bleeding or diarrhea (at least 4 stools per day over baseline); a positive GI biopsy is not sufficient to document clinical involvement
  * Autonomic nerve involvement is defined as orthostasis, symptoms of nausea or dysgeusia, gastric atony by gastric emptying scan, diarrhea, or constipation
  * Soft tissue and lymphatic involvement may be ascertained based on classic physical exam findings (macroglossia, shoulder pad sign, raccoon eyes, carpal tunnel syndrome, synovial enlargement, firm enlarged lymph nodes) or biopsy
* Ineligible for autologous stem cell transplantation with melphalan 200 mg/m^2 or refuses to undergo transplantation
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Amyloid cardiac biomarker stage I or II disease

  * The amyloid cardiac staging system is based on NT-proBNP and troponin-T levels. If troponin T (cTnT) is not available at local institution then troponin I (cTnI) may be used. Thresholds for cTnT, cTnI, and NT-proBNP are < 0.035 ug/L, < 0.1 ug/L, and < 332 ng/L, respectively. Stage I patients have both troponin-T (or I) and NT-proBNP below the threshold. Stage II patients have either troponin-T (I) or NT-proBNP above the threshold. Stage III patients have troponin-T (or I) and simultaneous NT-proBNP above the threshold. Stage III patients are further classified as "better risk" if NT-proBNP is over 332 ng/L but less than 6000 ng/L
* Negative pregnancy test
* Fertile patients must use effective contraception
* The absence of supine systolic blood pressure < 100 mmHg and difficult to manage symptomatic orthostatic hypotension
* Absolute neutrophil count (ANC) > 1,500/mm^3
* Platelet count > 140,000/mm^3
* Hemoglobin > 10 g/dL
* Total bilirubin < 2.5 mg/dL
* Alkaline phosphatase < 5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) < 3 times ULN
* Creatinine clearance > 30 mL/min
* Bone marrow plasma cells < 30%
* Human immunodeficiency virus (HIV)-positivity allowed provided the following criteria are met:

  * No history of acquired immunodeficiency syndrome (AIDS)-defining events including history of CD4 cell count < 200/mm^3
  * Current CD4 cell count >= 350/mm^3
  * Not receiving zidovudine or stavudine
  * No secondary amyloidosis
* More than 3 weeks since radiotherapy

  * Enrollment of subjects who require radiotherapy (which must be localized in field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy
* More than 14 days since prior and no concurrent participation in clinical trials with other investigational agents not included in this trial

Exclusion Criteria:

* Pregnant or nursing
* Clinically overt myeloma (hypercalcemia or lytic bone lesions)
* Prior chemotherapy or radiotherapy for the treatment of myeloma or systemic light-chain amyloidosis
* History of sustained ventricular tachycardias
* Cardiac syncope
* Uncompensated New York Heart Association (NYHA) class III or IV congestive heart failure
* Uncontrolled infection
* Active malignancy within the past 5 years except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or adequately treated stage I cancer currently in complete remission
* Serious medical or psychiatric illness likely to interfere with study participation, including recent myocardial infarction (within the past 6 months) or poorly controlled diabetes mellitus
* Hypersensitivity to bortezomib, boron, or mannitol
* Grade 2 or higher peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11-12 (Actual); Study Completion 2012-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dispenzieri, M.D., Study Chair — Mayo Clinic
Locations (209):
- United States (209):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Indiana University Medical Center, Indianapolis, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Union Hospital of Cecil County, Elkton, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Providence Hospital, Southfield, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - The Jewish Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Western Oncology Research Consortium, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazelton, Hazleton, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Columbia Basin Hematology and Oncology PLLC, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - D N Greenwald Center, Mukwonago, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital - ProHealth Care, Waukesha, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG member institutions between November 1, 2010 and September 7, 2012.
Period: Overall Study
Arm/Group | Arm A (Mel-Dex) | Arm B (B-Mel-Dex)
Started | 6 | 5
Completed | 5 | 3
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Mel-Dex) | Arm B (B-Mel-Dex) | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Median (Full Range); unit: years] | 68 [61 to 78] | 66 [44 to 72] | 67 [44 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Hematologic Overall Response (Partial Response [PR]+ Very Good PR [VGPR]+ Amyloid Complete Response [ACR]+ Stringent Complete Response [sCR]) After 3 Months (3 Cycles) of Therapy
Description: sCR: ACR and no clonal cells in bone marrow (BM) ACR: Negative serum/urine immunofixation (IF), <5% plasma cells in BM, and normal serum FLC ratio VGPR: 1. PR and any of the following; 2. serum/urine M-protein detectable by IF but not measurable (NM) on electrophoresis (EP); (3) ≥90% reduction in serum M-component and urine M-protein <100 mg/24 hr if baseline serum measurable; (4) urine M-component <100 mg/24 hr and NM serum M-protein on serum protein EP if baseline urine measurable; (5) ≥90% drop in the difference between involved and uninvolved FLC levels if only FLC measurable PR: (1) ≥50% drop of serum M-protein and 24-hr urinary M-protein drop by ≥90% or to <200 mg/24 hr if baseline serum/urine measurable; or (2) ≥50% drop of serum M-protein if only serum measurable at baseline; or (3) 24-hr urinary M-protein drop by ≥90% or to <200 mg/24 hr if baseline urine measurable; or (4) ≥ 50% drop in the difference between involved and uninvolved FLC if only FLC measu
Time Frame: Assessed at 3 months
Population: All enrolled patients are included in this analysis.
Measure: Number (90% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm A (Mel-Dex) | Arm B (B-Mel-Dex)
Number analyzed (Participants) | 6 | 5
Proportion of patients | 0.33 [0.06 to 0.73] | 0.60 [0.19 to 0.92]

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Arm/Group | Arm A (Mel-Dex) | Arm B (B-Mel-Dex)
Serious Adverse Events (participants affected / at risk) | 1/6 | 3/5
Other Adverse Events (participants affected / at risk) | 1/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Mel-Dex) (N=6) | Arm B (B-Mel-Dex) (N=5)
Fatigue (General disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
White blood cell decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Mel-Dex) (N=6) | Arm B (B-Mel-Dex) (N=5)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Fatigue (General disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less